CLINICAL TRIAL: NCT04482088
Title: Piloting an Enhanced Protocol of Occupational Therapy in an Equine Environment for Youth With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Hearts and Horses Therapeutic Riding Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-10140H
Record Dates: First submitted 2020-07-16; First posted 2020-07-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder
Keywords: occupational therapy; equine-assisted services; hippotherapy
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: All participants will receive 10 weeks of occupational therapy in a clinic, followed by occupational therapy in an equine environment
Masking Description: The occupational therapist that rates goal attainment will be blinded to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OTC & OTEE (Experimental): Every participant will receive 10 weeks of occupational therapy in a clinic environment (OTC) followed by 10 weeks of occupational therapy in an equine environment
  Interventions: Behavioral: Occupational Therapy in an Equine Environment; Behavioral: Occupational Therapy in a Clinic (OTC)

INTERVENTIONS:
Behavioral: Occupational Therapy in an Equine Environment — 10 weeks of occupational therapy in an equine environment aimed at improving individual goals related to self-regulation, social communication, and play
  Other Names: OTEE-HORSPLAY
Behavioral: Occupational Therapy in a Clinic (OTC) — 10 weeks of occupational therapy in a clinic aimed at improving individual goals related to self-regulation, social communication, and play

SUMMARY:
The purpose of this study is to learn about occupational therapy for youth with autism in a traditional clinic environment, and in an equine environment. 20 youth with autism will participate in 10 weeks of occupational therapy in a clinic environment, followed by 10 weeks of occupational therapy in an equine environment. Caregivers will complete online surveys about their child's behavior. Occupational therapists and other stakeholders will provide feedback about the interventions. The therapy sessions that involve horses will be videotaped, and a researcher will look at the behaviors of the horses involved in the intervention. We will use the results of this study to improve the quality of both interventions.

DETAILED DESCRIPTION:
The purpose of this study is to assess the feasibility, acceptability, and preliminary efficacy of occupational therapy in an equine environment (OTEE) for youth with autism. As a feasibility study, this study aims to accomplish several key development tasks. Specifically, this study aims to:

1. Create a safe, feasible, and manualized control group that controls for non-animal critical elements of the OTEE intervention
2. Assess welfare of the therapy horses that are integrated into the OTEE intervention
3. Enhance the OTEE manual by increasing standardization, while still allowing for individualization

Design. We will implement a longitudinal design, where caregivers will complete outcomes measures at 1)pre-test, 2) after their child participates in 10 weeks of occupational therapy in a clinic environment and 3) after 10 weeks of occupational therapy in an equine environment.

Participants. Youth with ASD will be screened for inclusion in a 2-part process that includes 1) an online survey and 2) virtual screening visit using Microsoft Teams. After completing 10 weeks of occupational therapy in a clinic environment, youth will then participate in an additional screening visit and re-evaluation for OTEE to ensure they a) are able to mount and ride a horse (with assistance) for 10 minutes while following safety rules, and b) meet all PATH Intl criteria for participation in equine-assisted services. Twenty youth with autism and their caregivers will be enrolled in the study. Occupational therapists that deliver the interventions and other stakeholders (i.e. program coordinators, etc.) will also be asked to be research participants.

Occupational Therapy Evaluation. Each youth and caregiver will participate in an occupational therapy evaluation at Temple Grandin Equine Center (or virtually, depending on COVID guidelines in 2021) that include an occupational profile, semi-structured interview, social skills checklist, and collaborative goal setting. Therapists and caregivers will jointly determine three goals for each youth with autism in the domains of self-regulation, social communication, or social play.

Occupational Therapy in a Clinic (Control Group). The occupational therapy in a clinic environment will occur at Temple Grandin Equine Center on CSU's foothills campus. We will recruit occupational therapists to deliver the intervention who a) are licensed and registered occupational therapists, and b) have at least 1-year of experience providing occupational therapy to youth with autism. Included therapists will receive 5 hours of training before each 10-week intervention session, as well as participate in 1-hour case conferences every other week throughout the 10 week intervention session.

Youth with autism will be paired into dyads based on social communication and self-regulation abilities. Dyads will attend 10 weekly 60-minute sessions of occupational therapy that follow a general structure: greeting, activities in a play room, parent debrief, and goodbyes. Therapists will design intervention activities based on the following critical elements: direct instruction of goal behavior; activities in the playroom that elicit the goal behavior; positive reinforcement of goal behaviors; use of behavioral techniques to scaffold goal performance.

Hearts and Horses Screening Visit and Re-evaluation. Each youth will attend an additional screening visit for the second portion of the study, to ensure they can safely ride a horse with assistance and meet all medical and behavioral standards set forth by PATH Intl for participation in equine-assisted services. Caregivers will be asked to bring the Hearts and Horse enrollment packet, that includes physician signature that the youth can ride a horse. Then, youth will ride a horse for 15 minutes. Finally, caregivers and youth will participate in re-evaluations with an occupational therapist, to update or set new goals for 10 weeks of OTEE.

OTEE Intervention (Intervention group). The OTEE intervention will occur at Hearts and Horses Therapeutic Riding Center. The occupational therapists who will deliver the intervention are licensed and registered, have completed training by the American Hippotherapy Association, are PATH Intl registered instructors, and have experience delivering occupational therapy in an equine environment to youth with autism. Included therapists will receive 5 hours of training before each 10-week intervention session, as well as participate in 1-hour case conferences every other week throughout the 10-week intervention session.

Youth with autism will be paired into dyads based on social communication and self-regulation abilities. Dyads will attend 10 weekly 60-minute sessions of OTEE. Sessions follow a general structure: greetings, activities with horses, parent debrief, goodbyes. Therapists design intervention activities based on these critical elements: a) incorporation of horses to optimize attention and engagement (includes use of equine movement to facilitate optimal arousal) b) direct instruction of goal behavior, c) activities with horses that elicit the goal behavior, d) positive reinforcement of goal behaviors, and e) use of behavioral techniques to scaffold goal performance.

Equine Welfare. OTEE sessions will be videotaped. Noldus software will be used to analyze equine behaviors using an applied ethogram, a behavioral scoring system in horses incorporated in equine-assisted services that determines the presence or absence of stress.

Fidelity. Dr. Peters will rate the fidelity of 25% of intervention and control sessions. Therapists will also provide self-ratings of fidelity for 20% of intervention and control sessions.

Outcome Measures. All youth/caregiver outcome measures will be collected three times: once before occupational therapy in a clinic environment, once before OTEE, and once after OTEE. Caregivers will be asked to complete online surveys that include the following assessments: Aberrant Behavior Checklist- Community (ABC-C) irritability and hyperactivity sub-scales, Social Responsiveness Scale Second Edition (SRS-2), Pediatric Evaluation of Disability Inventory Computer Adaptive Test for Autism Spectrum Disorders (PEDICAT-ASD), Emotional Dysregulation Inventory (EDI), and World Health Organization Quality of Life- Brief (WHOQOL-Brief). After each 10-week session, an occupational therapist blinded to treatment condition will call each caregiver and conduct a semi-structured interview in order to rate the child's performance on occupational performance goals using goal attainment scaling methods.

Therapists will be asked to fill out feedback forms every other week during case conferences, to gather immediate feedback on intervention delivery. After the evaluations/re-evaluations, therapists will be asked to complete a short survey about the feasibility and acceptability of the evaluations. At the conclusion of each 10-week session, therapists and other stakeholders (i.e. program coordinator, etc.) will be asked to complete short surveys about intervention acceptability, as well as attend a 1-hour audiotaped focus group to gather feedback on the intervention manual.

Data Analysis. To assess feasibility and acceptability, we will calculate rates of attendance, attrition, fidelity, assessment completion, safety events, and satisfaction. We will conduct content analysis of focus group and feedback form data to inform intervention and control manual revisions. Preliminary efficacy will be assessed using appropriate parametric or non-parametric statistics.

ELIGIBILITY:
Inclusion Criteria:

* Score ≥ 15 on the Social Communication Questionnaire
* Diagnosed with autism by a community provider
* Meet clinical cut-offs for autism on the ADOS or ADOS-2
* Can follow 1-step directions
* Score >10 on ABC-C irritability subscale
* Meet symptom criterion score of CASI-5 for mood, anxiety, or ADHD diagnosis
* Meet PATH Intl medical and behavioral standards, and can ride a horse for 10 minutes while following safety rules.

Exclusion Criteria:

* Participated in equine-assisted activities or therapies for 5 or more hours in the last 6 months
* Weigh more than 200 pounds

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Change in Goal Performance using Goal Attainment Scaling | 10 weeks
  Performance on individualized occupational performance goals

SECONDARY OUTCOMES:
Change in Aberrant Behavior Checklist- Community | 10 weeks
  Irritability and hyperactivity
Change in Social Responsiveness Scale, Second Edition | 10 weeks
  Social Functioning
Change in Pediatric Disability Inventory Computer Adaptive Test for Autism Spectrum Disorders | 10 weeks
  Adaptive behaviors
Change in World Health Organization Quality of Life- BREF | 10 weeks
  Quality of Life
Change in Emotional Dysregulation Inventory | 10 weeks
  Emotional Regulation

CONTACTS AND LOCATIONS:
Locations (1):
- Temple Grandin Equine Center Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Temple Grandin Equine Center — http://tgec.agsci.colostate.edu/